CLINICAL TRIAL: NCT02836041
Title: A Pilot Study: Sleep in Hospitalized Children With Cancer and Related Diseases
Brief Title: Sleep in Hospitalized Children at MSKCC
Status: Completed | Type: Observational
Sponsor: Memorial Sloan Kettering Cancer Center (Other)
Collaborators: Johns Hopkins University (Other); Weill Medical College of Cornell University (Other)
Responsible Party: Sponsor
Other Study IDs: 16-866
Record Dates: First submitted 2016-07-14; First posted 2016-07-18 (Estimated); Last update posted 2021-05-28 (Actual); Status verified 2021-05

CONDITIONS: Pediatric Cancer Patients
Keywords: assess sleep; Sleep Deprivation; 16-866
MeSH Terms: conditions — Sleep Deprivation | interventions — Surveys and Questionnaires

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective

GROUPS / COHORTS (1):
- Pediatrics cancer patients: Eligible patients will be approached for enrollment after their first night in the hospital (i.e.: not on day of admission). Patient/parent will be asked to complete a brief questionnaire describing the child's general sleep habits prior to admission. The parent and/or child will then be asked to complete a questionnaire describing sleep while in the hospital; this in-hospital sleep questionnaire will be obtained for 3 consecutive nights after enrollment, or until discharge, whichever is soonest. A subgroup of patients (between the ages of 5 and 18) will be invited to participate in an additional aspect of the study, where they wear an actigraph (a small device that looks like a watch) for up to 72 hours. This device reliably measures sleep by monitoring the child's motion. This will be used to relate sleep perception to more objective measures of sleep as provided by actigraphy.
  Interventions: Behavioral: questionnaires; Device: actigraph

INTERVENTIONS:
Behavioral: questionnaires — Pre-hospital sleep questionnaire completed (Brief Infant Sleep Questionnaire (BISQ)7 in children 0-3 years old; Children's Sleep Habits Questionnaire (CSHQ)8 in children 4 years and older). Subsequent Day(s):
  In-hospital sleep questionnaire completed between one and three times per subject (Sleep at MSK questionnaire (SAM), adapted from Sleep in a Children's Hospital (SinCH)9 by Dr. Lisa Meltzer). (Patients will be observed for up to 3 consecutive nights in total).
Device: actigraph — This device reliably measures sleep by monitoring the child's motion.

SUMMARY:
The investigators want to better understand how children sleep at night at MSKCC, so that the investigators can learn how to improve the sleeping environment.

ELIGIBILITY:
Inclusion Criteria:

* Parent/Patient must provide written consent
* Patient must be between the ages of: Newborn - ≤ 18 years of age
* Patient is expected to be admitted to the Pediatric floor at MSK for at least 2 nights (patients/parents will not be approached for consent on day of admission or day of discharge)
* Patient/parent must be English speaking

Exclusion Criteria:

* Expected length of stay of fewer than 2 nights (for example.: if admitted Monday and discharged Tuesday, patient/parent will not be eligible).
* Patient /Parent unable to complete questionnaire due to education or language barriers.
* Patients admitted to the PICU. (Only children on M9 will be included. It is known that sleep in the PICU is highly disordered; as such, we will be excluding PICU patients from this study).

Ages: 0 Months to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: All eligible patients admitted to the pediatric floor at MSK.
Sampling Method: Non-Probability Sample
Enrollment: 66 (Actual)
Dates: Start 2016-07-07 (Actual); Primary Completion 2021-05-26 (Actual); Study Completion 2021-05-26 (Actual)

PRIMARY OUTCOMES:
quality of sleep | 3 nights
  (using the Sleep at MSK questionnaire)

CONTACTS AND LOCATIONS:
Overall Officials: Chani Traube, MD, Principal Investigator — Memorial Sloan Kettering Cancer Center
Locations (1):
- Memorial Sloan Kettering Cancer Center, New York, New York, United States

REFERENCES:
- See also: Memorial Sloan Kettering Cancer Center — https://www.mskcc.org/